CLINICAL TRIAL: NCT02813928
Title: Diagnostic and Prognosis Value of Circulating DNA for CRC Patients' Surveillance After Curative Treatment
Acronym: ADNCirc
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Limoges (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: I15031
Record Dates: First submitted 2016-06-23; First posted 2016-06-27 (Estimated); Last update posted 2022-08-02 (Actual); Status verified 2022-06

CONDITIONS: Colorectal Cancer
Keywords: ColoRectal Cancer; Cancerology; Translational Research; ccfDNA
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ccfDNA analysis (Experimental): The level of circulating ccfDNA, defined as extra cellular DNA, increases in CRC patients. The Inplex® method could validate the use of ccfDNA as a cancer biomarker in terms of prognosis and surveillance.
  Interventions: Genetic: ccfDNA analysis

INTERVENTIONS:
Genetic: ccfDNA analysis — The level of circulating ccfDNA, defined as extra cellular DNA, increases in CRC patients. The Inplex® method could validate the use of ccfDNA as a cancer biomarker in terms of prognosis and surveillance

SUMMARY:
Inspite of curative treatment 30-50% patients with ColoRectal Cancer (CRC) develop tumor relapse during the first 3 years after treatment of the primary tumor. Treatment of relapses is based on surgical resection, when possible, chemotherapy and targeted therapies. To detect recurrences or metastases, a surveillance strategy is recommended for patients able to withstand complementary treatment during a five-year period. Over this period, the probability of one false-positive result is 87%. Considering that less than 10% of recurrent patients are suitable for potentially curative treatment and that more intensive programs enable an increase of the overall rate of curative resection but do not result in reduced mortality, less time and cost-consuming, tailored follow-up is necessary. The level of circulating ccfDNA, defined as extra cellular DNA, increases in CRC patients. The Inplex® method could validate the use of ccfDNA as a cancer biomarker in terms of prognosis and surveillance.

Tubes for ccfDNA analysis will be taken during medical examination at the same time of the CEA dosage (if it was not made before the consultation). Cryotubes of plasma will be sent for analysis in the laboratory INSERM (National Health Institute) of Montpellier and the remaining plasma will be kept in biological collection.

Patients will have a consultation of follow-up every 3-4 months during which the dosage of CEA and ccfDNA will be realized as well as a medical examination, a general examination (weight, size, and blood pressure), an evaluation of the indices of performance status and a nutritional evaluation in case of loss of weight.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Primary diagnosis of stages II and III CRC:
* is already operated and histological proven (biopsy at least)
* is patient that must be operated: curative treatment for stages II and III CRC
* Patient benefiting from a program personalized by care
* Written informed consent

Exclusion Criteria:

* Patient already treated for stages II and III CRC and in surveillance
* Patient with indication or with palliative treatment
* Pregnant or nursing patients
* Known pregnancy
* Difficulties to understand the protocol
* Patients under protection measure (guardianship, curatorship, protection of justice)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 473 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2021-12 (Actual); Study Completion 2022-07 (Actual)

PRIMARY OUTCOMES:
The presence of recurrences detected for patients curatively treated for a CRC stages II and III within the 3 years of follow-up. | 3 years

CONTACTS AND LOCATIONS:
Locations (19):
- France (19):
  - Aurillac Hospital, Aurillac
  - Bergonie institute, Bordeaux
  - Bordeaux University Hospital, Bordeaux
  - Les Cèdres clinical, Brive-la-Gaillarde
  - Brive Hospital, Brivé
  - Cahors Hospital, Cahors
  - Clermont Ferrand University Hospital, Clermont-Ferrand
  - Gueret Hospital, Guéret
  - La marche clinical, Guéret
  - Limoges Hospital, Limoges
  - Montpellier Institute, Montpellier
  - Montpellier University Hospital, Montpellier
  - Moulins Hospital, Moulins
  - Saint Antoine AP-HP, Paris
  - Perigueux clinical, Périgueux
  - Périgueux Hospital, Périgueux
  - Saint Junien Hospital, Saint-Junien
  - Sainte feyre Hospital, Sainte-Feyre
  - Vichy Hospital, Vichy

IPD SHARING:
Plan to Share IPD: No
the data are anonymized